CLINICAL TRIAL: NCT03442218
Title: Use fo Antiseptic Solution for Vaginal Wash Before Cesarean Section in Patients With Premature Rupture of Membranes. A Randomized, Double Blind, Controlled Trial.
Brief Title: Use of Antiseptic Solution for Vaginal Wash Before Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Collaborators: Sistema Nacional de Investigación (SNI) - Panamá (Unknown)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Head - Research Department, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MHST2014-20
Record Dates: First submitted 2018-02-13; First posted 2018-02-22 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Operation Wound; Infection; Endometritis
Keywords: Cesarean; Operative site infection; Vaginal wash; Clorhexidine; Endometritis
MeSH Terms: conditions — Surgical Wound Infection; Endometritis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clorhexidine (Experimental): Vaginal wash with clorhexidine solution
  Interventions: Drug: Clorhexidine
- Saline solution (Placebo Comparator): Vaginal wash with saline solution
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Clorhexidine — Vaginal wash with clorhexidine solution previous to cesarean section in patients with premature rupture of membranes.
  Arms: Clorhexidine
Drug: Saline solution — Vaginal wash with saline solution previous to cesarean section in patients with premature rupture of membranes.
  Arms: Saline solution

SUMMARY:
To evaluate the rate of infections after cesarean sections in patients with premature rupture of membranes after vaginal wash either with an antiseptic solution (clorhexidine solution) vs. saline solution (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Women with gestation between 34 and 41 6/7 weeks.
* Premature rupture of membranes (> 6 hours).
* Use of prophylactic antibiotic 1 hour previous to cesarean section.

Exclusion Criteria:

* Any source of infection diagnosed previous to surgery.
* Fever of unknown origin previous to surgery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Number of cases of endometritis after cesarean section | 15 days
  Endometritis

SECONDARY OUTCOMES:
Number of cases of cesarean site infection | 15 days
  Operative site infection
Number of cases of fever (38°C or above) in the puerperium | 15 days
  Puerperal fever

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Panama

REFERENCES:
- [Derived] Urena N, Reyes O. Preoperative vaginal cleansing with chlorhexidine vs placebo in patients with rupture of membranes: a prospective, randomized, double-blind, placebo-control study. Am J Obstet Gynecol MFM. 2022 Mar;4(2):100572. doi: 10.1016/j.ajogmf.2022.100572. Epub 2022 Jan 17. PMID 35051671
- [Derived] Haas DM, Morgan S, Contreras K, Kimball S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2020 Apr 26;4(4):CD007892. doi: 10.1002/14651858.CD007892.pub7. PMID 32335895